CLINICAL TRIAL: NCT06265103
Title: Epilepsy Learning Healthcare System (ELHS) for Quality Care & Outcome Improvement
Brief Title: Epilepsy Learning Healthcare System (ELHS)
Acronym: ELHS
Status: Recruiting | Type: Observational
Sponsor: Epilepsy Foundation of America (Other)
Responsible Party: Sponsor
Other Study IDs: 20190407
Record Dates: First submitted 2020-05-28; First posted 2024-02-20 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Epilepsy; Seizure Disorder; Neurologic Disorder; Rare Diseases
Keywords: Focal seizures; Generalized seizures; Brain conditions; Developmental disorders; Rare diseases; Chronic condition; Health disparity; Seizure; Post-traumatic epilepsy (PTE); Post-stroke epilepsy
MeSH Terms: conditions — Epilepsy; Nervous System Diseases; Rare Diseases; Seizures; Brain Diseases; Developmental Disabilities; Chronic Disease; Epilepsy, Post-Traumatic | interventions — Quality Improvement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (12):
- Barrow Neurological Institute Comprehensive Epilepsy Center: Centers participating in ELHS will work towards accomplishing the improved process and clinical outcomes by implementing changes via Quality Improvement methodology in the context of a Chronic Care model. Specifically, programs will introduce common data elements and standardized epilepsy care metrics followed by rapid cycle feedback via site specific and overall network outcomes. Interventions will then be introduced based upon evidence-based recommendations to improve outcomes. Network-based changes to practice such as those suggested have never been realized in the domain of epilepsy to date.
  Interventions: Other: Clinical care and quality improvement
- Cincinnati Children's Hospital Medical Center: Centers participating in ELHS will work towards accomplishing the improved process and clinical outcomes by implementing changes via Quality Improvement methodology in the context of a Chronic Care model. Specifically, programs will introduce common data elements and standardized epilepsy care metrics followed by rapid cycle feedback via site specific and overall network outcomes. Interventions will then be introduced based upon evidence-based recommendations to improve outcomes. Network-based changes to practice such as those suggested have never been realized in the domain of epilepsy to date.
  Interventions: Other: Clinical care and quality improvement
- Children's Hospital of Philadelphia (CHOP): Centers participating in ELHS will work towards accomplishing the improved process and clinical outcomes by implementing changes via Quality Improvement methodology in the context of a Chronic Care model. Specifically, programs will introduce common data elements and standardized epilepsy care metrics followed by rapid cycle feedback via site specific and overall network outcomes. Interventions will then be introduced based upon evidence-based recommendations to improve outcomes. Network-based changes to practice such as those suggested have never been realized in the domain of epilepsy to date.
  Interventions: Other: Clinical care and quality improvement
- Children's Hospital of Orange County (CHOC): Centers participating in ELHS will work towards accomplishing the improved process and clinical outcomes by implementing changes via Quality Improvement methodology in the context of a Chronic Care model. Specifically, programs will introduce common data elements and standardized epilepsy care metrics followed by rapid cycle feedback via site specific and overall network outcomes. Interventions will then be introduced based upon evidence-based recommendations to improve outcomes. Network-based changes to practice such as those suggested have never been realized in the domain of epilepsy to date.
  Interventions: Other: Clinical care and quality improvement
- Mass General Hospital: Centers participating in ELHS will work towards accomplishing the improved process and clinical outcomes by implementing changes via Quality Improvement methodology in the context of a Chronic Care model. Specifically, programs will introduce common data elements and standardized epilepsy care metrics followed by rapid cycle feedback via site specific and overall network outcomes. Interventions will then be introduced based upon evidence-based recommendations to improve outcomes. Network-based changes to practice such as those suggested have never been realized in the domain of epilepsy to date.
  Interventions: Other: Clinical care and quality improvement
- Penn State Hershey: Centers participating in ELHS will work towards accomplishing the improved process and clinical outcomes by implementing changes via Quality Improvement methodology in the context of a Chronic Care model. Specifically, programs will introduce common data elements and standardized epilepsy care metrics followed by rapid cycle feedback via site specific and overall network outcomes. Interventions will then be introduced based upon evidence-based recommendations to improve outcomes. Network-based changes to practice such as those suggested have never been realized in the domain of epilepsy to date.
  Interventions: Other: Clinical care and quality improvement
- University of Cincinnati Gardner Neuroscience Institute: Centers participating in ELHS will work towards accomplishing the improved process and clinical outcomes by implementing changes via Quality Improvement methodology in the context of a Chronic Care model. Specifically, programs will introduce common data elements and standardized epilepsy care metrics followed by rapid cycle feedback via site specific and overall network outcomes. Interventions will then be introduced based upon evidence-based recommendations to improve outcomes. Network-based changes to practice such as those suggested have never been realized in the domain of epilepsy to date.
  Interventions: Other: Clinical care and quality improvement
- University of Southern California (USC): Centers participating in ELHS will work towards accomplishing the improved process and clinical outcomes by implementing changes via Quality Improvement methodology in the context of a Chronic Care model. Specifically, programs will introduce common data elements and standardized epilepsy care metrics followed by rapid cycle feedback via site specific and overall network outcomes. Interventions will then be introduced based upon evidence-based recommendations to improve outcomes. Network-based changes to practice such as those suggested have never been realized in the domain of epilepsy to date.
  Interventions: Other: Clinical care and quality improvement
- UT Southwestern Children's Dallas: Centers participating in ELHS will work towards accomplishing the improved process and clinical outcomes by implementing changes via Quality Improvement methodology in the context of a Chronic Care model. Specifically, programs will introduce common data elements and standardized epilepsy care metrics followed by rapid cycle feedback via site specific and overall network outcomes. Interventions will then be introduced based upon evidence-based recommendations to improve outcomes. Network-based changes to practice such as those suggested have never been realized in the domain of epilepsy to date.
  Interventions: Other: Clinical care and quality improvement
- Brigham & Women's Hospital: Centers participating in ELHS will work towards accomplishing the improved process and clinical outcomes by implementing changes via Quality Improvement methodology in the context of a Chronic Care model. Specifically, programs will introduce common data elements and standardized epilepsy care metrics followed by rapid cycle feedback via site specific and overall network outcomes. Interventions will then be introduced based upon evidence-based recommendations to improve outcomes. Network-based changes to practice such as those suggested have never been realized in the domain of epilepsy to date.
  Interventions: Other: Clinical care and quality improvement
- Children's Hospital Los Angeles: Centers participating in ELHS will work towards accomplishing the improved process and clinical outcomes by implementing changes via Quality Improvement methodology in the context of a Chronic Care model. Specifically, programs will introduce common data elements and standardized epilepsy care metrics followed by rapid cycle feedback via site specific and overall network outcomes. Interventions will then be introduced based upon evidence-based recommendations to improve outcomes. Network-based changes to practice such as those suggested have never been realized in the domain of epilepsy to date.
  Interventions: Other: Clinical care and quality improvement
- University of Colorado Anshutz: Centers participating in ELHS will work towards accomplishing the improved process and clinical outcomes by implementing changes via Quality Improvement methodology in the context of a Chronic Care model. Specifically, programs will introduce common data elements and standardized epilepsy care metrics followed by rapid cycle feedback via site specific and overall network outcomes. Interventions will then be introduced based upon evidence-based recommendations to improve outcomes. Network-based changes to practice such as those suggested have never been realized in the domain of epilepsy to date.
  Interventions: Other: Clinical care and quality improvement

INTERVENTIONS:
Other: Clinical care and quality improvement — All eligible patients at each center will be included in the registry for clinical care, quality improvement and other activities that do not meet the regulatory requirements of human subjects research. Use of data for these purposes is not considered to be a human subjects research activity and will be covered under a Business Associates Agreement and a Participation and Data Use Agreement.

SUMMARY:
The Epilepsy Learning Health System (ELHS) is a quality improvement and research network to improve outcomes for people with epilepsy. The ELHS is designed as a model of value-based chronic care for epilepsy as envisioned by the National Academies of Medicine Committee in their landmark reports "The Learning Health System" and "Epilepsy Across the Spectrum: Promoting Health and Understanding".

The ELHS network is a collaboration among clinicians, patients and researchers that promotes the use of data for multiple purposes including one-on-one clinical care, population management, quality improvement and research. The ELHS Registry includes data on children and adults with epilepsy collected during the process of standard epilepsy care. These data are used to create population health reports and to track changes in outcomes over time. ELHS teams use quality improvement methods, such as Plan-Do-Study-Act (PDSA) cycles, to continuously learn how to improve care.

DETAILED DESCRIPTION:
The Epilepsy Learning Healthcare System (ELHS; pronounced el-is) involves patients and families living with epilepsy, clinicians who provide epilepsy care (including pediatric and adult epileptologists, neurology nurses, and others), community services providers, as well as researchers with clinical research expertise in community-based, observational, interventional, implementation and dissemination studies. Each stakeholder agrees to work together to improve outcomes for people with epilepsy.

NETWORK AIM The purpose of the network is to improve seizure control and quality of life for people with epilepsy through a learning healthcare system, in which clinical data are collected, analyzed, and rapidly disseminated to change practice.

BACKGROUND Epilepsy is a chronic neurological disorder characterized by unprovoked seizures. Epidemiological data indicate that 10% of Americans will suffer at least one seizure at some point in their lives, and 1-2% of Americans have epilepsy. Active epilepsy affects 3.4 million Americans - currently estimated at 2.9 Million adults and around 460,000 children. At least 50% of the total population of individuals with epilepsy will have started having seizures at less than 20 years of age. More than half of U.S. adults with active epilepsy have high school diploma/GED or less education. Compared to the general public, people with epilepsy have higher rates of premature mortality, injury, cognitive impairment, depression, social isolation, and unemployment. In addition, there are health disparities (HD) in epilepsy that create worse health outcomes for individuals belonging to race/ethnicity minority groups or low-income households, those living in rural areas, and individuals with opposite or non-binary gender preferences. Epilepsy disparities result in worse mental health, more frequent emergency department visits, increased hospitalization rates, and increased risk of early death for these underserved groups.

Epilepsy is not a single disease. Rather, it is a heterogeneous set of disorders with genetic and acquired etiologies. The diversity of seizure types, epilepsy syndromes, outcomes and etiologies, cannot be overstated. It is likely that the extreme heterogeneity of the epilepsies is at least partially responsible for slow progress towards meaningful treatment strategies to improve outcomes. For some, epilepsy is a manageable chronic illness -- affected individuals have risen to the highest echelons of professional success. However, for others, epilepsy is a devastating and progressive disease leading to cognitive regression and early death. Wide variations in epilepsy care delivery and clinical practice may also contribute to poor individual outcomes.

The ELHS community will work towards its mission of improving outcomes for children and adults with Epilepsy by setting up a platform to support continuous and sustained improvement activities.

The ELHS network uses the Institute for Healthcare Improvement's "Model for Improvement", focusing on the three questions - What are we trying to accomplish? How will we know that a change is an improvement? What change can we make that will result in improvement? Iterative Plan- Do-Study-Act (PDSA) learning cycles are used to test and implement changes. The Model for Improvement is widely accepted across healthcare systems as a method to improve quality and health outcomes. It is used successfully in a growing number of patient safety and disease-focused learning health networks.

With guidance from experts in QI and care delivery, participating programs collect and share data, test specific changes in care, and determine how to redesign and incorporate improvements into daily practice. Most measures are reported monthly and shared transparently across the ELHS Network to generate discussion and drive QI efforts. Network-wide data are reviewed monthly on Action Period calls to learn from the variation amongst programs and to recognize and celebrate network-wide improvements.

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible to participate in this registry-based study, an individual must meet all of the following criteria:

  * Patient is in an established care relationship with the ELHS site

Exclusion Criteria:

* An individual who meets any of the following criteria will be excluded from participation in this registry-based research study:

  * Patients who are not currently in nor expect to be in an established care relationship with the ELHS site (for example, patients who are being seen at the center for a second opinion only).
  * Patients who do not, after diagnostic evaluation, meet criteria for a diagnosis of epilepsy will not be analyzed in epilepsy-specific population groups. However, these non-epilepsy patients will not be excluded from the registry.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People of all ages diagnosed with epilepsy by a physician and in an established care relationship, and their families and caregivers.
Sampling Method: Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2019-03-20 (Actual); Primary Completion 2099-02-14 (Estimated); Study Completion 2099-02-14 (Estimated)

PRIMARY OUTCOMES:
Seizure Frequency | 02/2099
  *Seizure frequency: A record of the number of seizures gathered from patient records, journal, or calendar OR the average or typical recent seizure frequency, often expressed as the average daily, weekly, or monthly seizure frequency since the last visit.
Seizure Freedom | 02/2099
  Percent of all patients with visits within the time interval who have had no seizures in the last 12 months. This is a population outcome metric.
Quality of Life documentation | 02/2099
  Percent of all visits at which a QOL assessment* is completed by the patient. This is a visit-based process metric.
Screening for Barriers to Medication Adherence | 02/2099
  Percent of all visits at which a Barriers to Medication Adherence Tool is completed by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Brandy Fureman, PhD, Principal Investigator — Epilepsy Foundation
Locations (13):
- United States (13):
  - Barrow Neurological Institute Comprehensive Epilepsy Center, Phoenix, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of Southern California, Los Angeles, California
  - UC Health University of Colorado Anshutz, Aurora, Colorado
  - Epilepsy Foundation, Bowie, Maryland
  - Partners - Massachusetts General Hospital Epilepsy Service (MGH)/ Partners - Brigham and Women's (BWH), Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital Comprehensive Epilepsy Center (CCHMC), Cincinnati, Ohio
  - University of Cincinnati Gardner Neuroscience Institute Epilepsy Center, Cincinnati, Ohio
  - Penn State Hershey, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia (CHOP), Philadelphia, Pennsylvania
  - UT Southwestern Children's Dallas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
To expand the possibilities for conducting outcomes research beyond the network investigators, data will be shared, following appropriate IRB review and approval prior to releasing data, with qualified investigators external to the network who are employed at, or affiliated with, institutions that are interested in conducting health services or comparative effectiveness research.
  Non-aggregate data must be maintained on an organization's secure servers and not downloaded to peripheral devices, including laptops, USB drives or workstations. Any individual or organization receiving the data must respect the limitations of the agreement including requirements on custody of data being maintained on organization servers.
Supporting Information: CSR
Time Frame: No time frame.
Access Criteria: External investigators and ELHS Participants may use shared data only under the terms of the agreement regardless of de-identification status. De-identification does not release data from terms of the agreement.
  Non-aggregate data must be maintained on an organization's secure servers and not downloaded to peripheral devices, including laptops, USB drives or workstations. Any individual or organization receiving the data must respect the limitations of the agreement including requirements on custody of data being maintained on organization servers.

REFERENCES:
- [Background] Fisher RS, Acevedo C, Arzimanoglou A, Bogacz A, Cross JH, Elger CE, Engel J Jr, Forsgren L, French JA, Glynn M, Hesdorffer DC, Lee BI, Mathern GW, Moshe SL, Perucca E, Scheffer IE, Tomson T, Watanabe M, Wiebe S. ILAE official report: a practical clinical definition of epilepsy. Epilepsia. 2014 Apr;55(4):475-82. doi: 10.1111/epi.12550. Epub 2014 Apr 14. PMID 24730690
- [Background] Zack MM, Kobau R. National and State Estimates of the Numbers of Adults and Children with Active Epilepsy - United States, 2015. MMWR Morb Mortal Wkly Rep. 2017 Aug 11;66(31):821-825. doi: 10.15585/mmwr.mm6631a1. PMID 28796763
- [Background] Institute of Medicine (US) Committee on the Public Health Dimensions of the Epilepsies; England MJ, Liverman CT, Schultz AM, Strawbridge LM, editors. Epilepsy Across the Spectrum: Promoting Health and Understanding. Washington (DC): National Academies Press (US); 2012. Available from http://www.ncbi.nlm.nih.gov/books/NBK91506/ PMID 22993876
- [Background] Thurman DJ, Logroscino G, Beghi E, Hauser WA, Hesdorffer DC, Newton CR, Scorza FA, Sander JW, Tomson T; Epidemiology Commission of the International League Against Epilepsy. The burden of premature mortality of epilepsy in high-income countries: A systematic review from the Mortality Task Force of the International League Against Epilepsy. Epilepsia. 2017 Jan;58(1):17-26. doi: 10.1111/epi.13604. Epub 2016 Nov 26. PMID 27888514
- [Background] Wasade VS, Spanaki M, Iyengar R, Barkley GL, Schultz L. AAN Epilepsy Quality Measures in clinical practice: a survey of neurologists. Epilepsy Behav. 2012 Aug;24(4):468-73. doi: 10.1016/j.yebeh.2012.05.017. Epub 2012 Jul 5. PMID 22770880
- [Background] Sanchez Fernandez I, Abend NS, Agadi S, An S, Arya R, Brenton JN, Carpenter JL, Chapman KE, Gaillard WD, Glauser TA, Goodkin HP, Kapur K, Mikati MA, Peariso K, Ream M, Riviello J Jr, Tasker RC, Loddenkemper T; Pediatric Status Epilepticus Research Group (pSERG). Time from convulsive status epilepticus onset to anticonvulsant administration in children. Neurology. 2015 Jun 9;84(23):2304-11. doi: 10.1212/WNL.0000000000001673. Epub 2015 May 6. PMID 25948729
- [Background] Mytinger JR, Joshi S; Pediatric Epilepsy Research Consortium, Section on Infantile Spasms. The current evaluation and treatment of infantile spasms among members of the Child Neurology Society. J Child Neurol. 2012 Oct;27(10):1289-94. doi: 10.1177/0883073812455692. Epub 2012 Aug 21. PMID 22914371
- [Background] Cui W, Kobau R, Zack MM; US Centers for Disease Control and Prevention, Epilepsy Program. Among adults with epilepsy reporting recent seizures, one of four on antiseizure medication and three of four not on medication had not seen a neurologist/epilepsy specialist within the last year, the 2010 and 2013 US National Health Interview Surveys. Epilepsy Behav. 2016 Aug;61:78-79. doi: 10.1016/j.yebeh.2016.04.031. Epub 2016 Jun 17. PMID 27318431
- [Background] Burneo JG, Jette N, Theodore W, Begley C, Parko K, Thurman DJ, Wiebe S; Task Force on Disparities in Epilepsy Care; North American Commission of the International League Against Epilepsy. Disparities in epilepsy: report of a systematic review by the North American Commission of the International League Against Epilepsy. Epilepsia. 2009 Oct;50(10):2285-95. doi: 10.1111/j.1528-1167.2009.02282.x. Epub 2009 Sep 3. PMID 19732134
- [Background] Faught E, Richman J, Martin R, Funkhouser E, Foushee R, Kratt P, Kim Y, Clements K, Cohen N, Adoboe D, Knowlton R, Pisu M. Incidence and prevalence of epilepsy among older U.S. Medicare beneficiaries. Neurology. 2012 Feb 14;78(7):448-53. doi: 10.1212/WNL.0b013e3182477edc. Epub 2012 Jan 18. PMID 22262750
- [Background] Avetisyan R, Cabral H, Montouris G, Jarrett K, Shapiro GD, Berlowitz DR, Kase CS, Kazis LE. Evaluating racial/ethnic variations in outpatient epilepsy care. Epilepsy Behav. 2013 Apr;27(1):95-101. doi: 10.1016/j.yebeh.2012.12.020. Epub 2013 Feb 9. PMID 23399943
- [Background] Jette N, Quan H, Faris P, Dean S, Li B, Fong A, Wiebe S. Health resource use in epilepsy: Significant disparities by age, gender, and aboriginal status. Epilepsia. 2008 Apr;49(4):586-93. doi: 10.1111/j.1528-1167.2007.01466.x. Epub 2007 Dec 28. PMID 18177361
- [Background] Schiltz NK, Koroukian SM, Singer ME, Love TE, Kaiboriboon K. Disparities in access to specialized epilepsy care. Epilepsy Res. 2013 Nov;107(1-2):172-80. doi: 10.1016/j.eplepsyres.2013.08.003. Epub 2013 Aug 16. PMID 24008077
- [Background] Sim Y, Nokes B, Byreddy S, Chong J, Coull BM, Labiner DM. Healthcare utilization of patients with epilepsy in Yuma County, Arizona: do disparities exist? Epilepsy Behav. 2014 Feb;31:307-11. doi: 10.1016/j.yebeh.2013.10.018. Epub 2013 Nov 5. PMID 24210458
- [Background] Institute of Medicine (US) Roundtable on Evidence-Based Medicine; Olsen L, Aisner D, McGinnis JM, editors. The Learning Healthcare System: Workshop Summary. Washington (DC): National Academies Press (US); 2007. Available from http://www.ncbi.nlm.nih.gov/books/NBK53494/ PMID 21452449
- [Background] Jeste DV, Palmer BW, Appelbaum PS, Golshan S, Glorioso D, Dunn LB, Kim K, Meeks T, Kraemer HC. A new brief instrument for assessing decisional capacity for clinical research. Arch Gen Psychiatry. 2007 Aug;64(8):966-74. doi: 10.1001/archpsyc.64.8.966. PMID 17679641